CLINICAL TRIAL: NCT01466738
Title: Clinical Characterization of a Human Rhinovirus Type 16 Challenge Pool Following Intranasal Administration to Healthy Adult Subjects
Brief Title: A Study of Human Rhinovirus Type 16 (HRV-16) Following Administration in the Nose of Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centocor Ortho Biotech Services, L.L.C. (Industry)
Responsible Party: Sr. Director, Translational Medicine, Janssen Research and Development, US
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CR018733; NOCOMPOUNDASH1001 (Other: Centocor Ortho Biotech Services, L.L.C.)
Record Dates: First submitted 2011-11-04; First posted 2011-11-08 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: Healthy volunteer; Rhinovirus; Cold virus; HRV-16

ARMS (2):
- HRV-16 (100 TCID50) (Experimental)
  Interventions: Biological: HRV-16 (100 TCID50)
- HRV-16 (1000 TCID50) (Experimental)
  Interventions: Biological: HRV-16 (1000 TCID50)

INTERVENTIONS:
Biological: HRV-16 (100 TCID50) — Each volunteer will receive a single administration of 100 TCID50 of HRV-16 in a total volume of approximately 1.0 mL administered via 4 intranasal instillations.
  Arms: HRV-16 (100 TCID50)
Biological: HRV-16 (1000 TCID50) — Each volunteer will receive a single administration of 1000 TCID50 of HRV-16 in a total volume of approximately 1.0 mL administered via 4 intranasal instillations.
  Arms: HRV-16 (1000 TCID50)

SUMMARY:
The purpose of this study is to evaluate the safety and clinical characteristics of a quantity of human rhinovirus Type 16 (HRV-16) in healthy volunteers. This source of HRV-16 will be subsequently used in viral challenge studies with new compounds that are intended to treat respiratory diseases.

DETAILED DESCRIPTION:
This is an open-label study in which all participants know the investigational substance being tested. Participants will be inoculated in the nose with HRV-16 and evaluated for the occurrence of cold symptoms and other indicators. There will be 3 phases: a screening phase, an HRV-16 infection phase, and a follow-up phase. The dose of virus being tested in this study has been previously used in other challenge studies. The total length of participation in the study will be about 4 weeks. Participant safety will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrate an understanding of the study and sign an informed consent form prior to any study-related procedures
* Healthy with no clinically significant abnormalities as determined by medical history
* Women must be neither pregnant nor lactating (producing breast milk) and have a negative urine pregnancy test at Screening Visit 1
* Women of child-bearing potential and all men must agree to use adequate birth control measures (as determined by the investigator) and must agree to continue to use such measures and not plan a pregnancy until after the Day 6 visit
* Men must agree not to donate sperm during the study through the Day 6 visit

Exclusion Criteria:

* Have a documented serum-neutralizing antibody titer of > 2-fold dilution to HRV-16 in the blood sample within approximately 40 days of Screening Visit 2
* Live with a family member who cares for the elderly, infants, or small children (eg, nursing home or day care provider), or live with someone who has a chronic lung disease, premature infant, or immunocompromised individual
* Require a prescription or over-the-counter medication on a regular basis (3 or more times per week), except contraceptive preparations, hormone replacement therapy, or topical acne medication
* Have a history of chronic disease that the Investigator believes are clinically significant
* Have a history of chronic headaches (eg frequent migraines, cluster headaches) with 3 or more headaches per week

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Clinical symptoms to HRV-16 | 6 days
  Clinical symptoms to HRV-16 will be assessed using the Cold Symptom Assessment form, which is a 5-point scale of the severity of cold symptoms.
Serological Response | Approximately 4 weeks
  Blood samples will be evaluated for serum-neutralizing antibody titer levels to HRV-16.

SECONDARY OUTCOMES:
The number of adverse events | Approximately 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Centocor Ortho Biotech Services, L.L.C. Clinical Trial, Study Director — Centocor Ortho Biotech Services, L.L.C.
Locations (1):
- Charlottesville, Virginia, United States